CLINICAL TRIAL: NCT03064464
Title: Community-associated Staphylococcus Aureus Infections in China: Epidemiology, Molecular Characteristics, Treatment, and Outcome
Brief Title: CA-MRSA Infection in China: Epidemiology, Molecular Characteristics, Treatment, and Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Jian-cang Zhou M.D., Department of Infectious Diseases, Sir Run Run Shaw Hospital
Other Study IDs: SRRSH-MRSA01
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Community-Acquired Infections; Methicillin-resistant Staphylococcus Aureus
Keywords: methicillin-resistant Staphylococcus aureus
MeSH Terms: conditions — Community-Acquired Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bacterial isolates
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CA-MRSA infection: None intervention
  Interventions: Other: None Intervention
- HA-MRSA infection: None intervention
  Interventions: Other: None Intervention
- CA-MSSA infection: None intervention
  Interventions: Other: None Intervention

INTERVENTIONS:
Other: None Intervention — It is observational study, no interventios to any of the three study arms

SUMMARY:
Community-associated methicillin-resistant Staphylococcus aureus (CA-MRSA), strains of MRSA that are able to infect otherwise healthy people outside of hospital settings, emerged in the late 1990s and have recently arisen in many countries around the globe. CA-MRSA strains are usually distinguished from their HA-MRSA counterparts by the following characteristics: Firstly, CA-MRSA strains are usually susceptible to non-lactam antibiotics. Secondly, CA-MRSA harbors type IV and V SCCmec elements, which are shorter than the traditional type I, II, and III SCCmec elements found in HA-MRSA strains. Thirdly, certain successful clones are associated with outbreaks of CA-MRSA infections reported in specific geographical locations. For example, ST1 and ST8 isolates are mostly reported in the USA and Canada, ST80 isolates are commonly found in Europe, and ST59 isolates are encountered in the Asia-Pacific region. Notably, all these characteristics have substantial limitations for discriminating CA-MRSA isolates due to their complex backgrounds. Although there were more and more studies of CA-MRSA in European countries and the US, few national epidemiological data were available about China. In this study, we investigated the epidemiological, clinical and molecular characteristics of CA-MRSA isolates recovered in Chinese hospitals, in order to understand the changing epidemiology of MRSA in China.

DETAILED DESCRIPTION:
Eligibility criteria:

1. Inclusion criteria: Patients (Child, Adult) with infections caused by S. aureus from the sites as follows: blood stream, skin or soft tissue, cerebrospinal fluid, bone and joint, genitourinary tract, infection of indwelling intravascular device, surgical wound, respiratory tract (organism grown from sputum and infiltrate on chest X-ray), peritoneal fluid or other otherwise sterile body fluids.
2. Exclusion criteria: Patients with S. aureus from anterior nares or throat swabs cultures (colonization).

Outcome measures:

1. Community-associated methicillin-resistant Staphylococcus aureus (CA-MRSA) infection rates in patients with S. aureus infections in Chinese hospitals.
2. Risk factors and clinical outcomes of CA-MRSA infection
3. Molecular characteristics of CA-MRSA isolates recovered in Chinese hospitals.

Definition:

A MRSA infection was considered to be HA-MRSA by the CDC epidemiologic definitions if, in the year prior to culture, the subject had surgery, hospitalization, hemodialysis or a stay in a long-term care facility, if an indwelling vascular catheter was in place at the time of culture, or if the subject was an inpatient hospitalized for 2 days at the time of culture. Otherwise, the subject was considered to have a CA-MRSA infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients (Child, Adult) with infections caused by S. aureus from the sites as follows: blood stream, skin or soft tissue, cerebrospinal fluid, bone and joint, genitourinary tract, infection of indwelling intravascular device, surgical wound, respiratory tract (organism grown from sputum and infiltrate on chest X-ray), peritoneal fluid or other otherwise sterile body fluids.

Exclusion Criteria:

* Patients with S. aureus from anterior nares or throat swabs cultures for colonization screening purpose.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All child and adult patients with Staphylococcus aureus visited any of the 60 particitant hospitals during the study period were included.
Sampling Method: Non-Probability Sample
Enrollment: 5400 (Estimated)
Dates: Start 2016-12-15 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of CA-MRSA infections in China | During the study period (Two years)
  Community-associated methicillin-resistant Staphylococcus aureus (CA-MRSA) infection rates in patients with S. aureus infections in Chinese hospitals

SECONDARY OUTCOMES:
Clonal Distribution of CA-MRSA in China | During the study period (Two years)
  The distribution of sequence types in CA-MRSA isolates from China

CONTACTS AND LOCATIONS:
Overall Officials: Yun-song Yu, MD, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided